CLINICAL TRIAL: NCT02735655
Title: The Global Status and the Unmet Needs for Training in Endoscopy; a World Endoscopy Organization Web Based Survey
Brief Title: Global State of Digestive Endoscopy Training Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Lecturer of Internal Medicine, Al-Azhar University
Other Study IDs: WEO-ES-1
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Gastrointestinal Endoscopy Training
Keywords: endoscopy; Education; capsule endoscopy; Cholangiopancreatography, Endoscopic Retrograde; esophagogastroduodenoscopy; colonoscopy; Double-Balloon Enteroscopy; Global status; unmet need

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Physician's opinion — To get physician's opinion about the current global state of gastrointestinal endoscopy training programs and to identify the unmet needs and how to improve it through a web based questionnaire.

SUMMARY:
This is a 10 minutes web based survey aims at exploring the current, global state of digestive endoscopy training among physicians to identify what are the unmet needs and how to improve it.

DETAILED DESCRIPTION:
Currently, gastrointestinal (GI) endoscopy training is not a standardized and is variable from country to country. A number of certifying authorities in different countries grant privileges of performing GI endoscopy according to predefined rules, requisites and regulations, especially in the Western countries (1-4). However, in many other countries, physicians who perform GI endoscopy as part of their medical practice may not require to be certified or acknowledged by a relevant regulatory body (5-8).

In the absence of quality assessment of GI training, patient safety and evidence-based medical care cannot be guaranteed. According to major societies of GI endoscopy, the credentialing decisions for GI endoscopy should be based on the evaluation of physicians' qualifications and procedural skills, as assessed by experienced doctors with whom they have trained, not solely on a simple counting of procedures performed (9). Therefore, there is a need for a WEO training guideline that defines training duration, procedural skills and competency that should be acquired by young GI endoscopists during their endoscopy training.

It is particularly important for WEO to standardize the fundamentals of GI endoscopy training globally by developing recommendations on endoscopic education and training to help medical institutions ensure the technical and cognitive competence of individuals requesting endoscopic privileges.

Objective:

To assess the current global state of GI endoscopy training programs and to identify the unmet needs and how to improve it through a web based questionnaire.

Methods:

Endoscopists from all over the world will be invited to answer in the questionnaire through e-mail invitations. Results will be analyzed to assess the current global status of GI endoscopy training in their countries, the unmet needs and to how improve it.

Survey link:

http://www.surveymonkey.net/create/survey/preview?r=true&sm=R74C8rWWwbO8_2BQM2fg9Yr5HcAtrkz8XwZogb4Bbaqr8oC9mFJrq8WAvNY33O45r1

ELIGIBILITY:
Inclusion Criteria:

* Physicians practicing gastrointestinal endoscopy from all over the world

Exclusion Criteria:

* Any other persons whom are not physicians or physicians not practicing gastrointestinal endoscopy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians practicing gastrointestinal endoscopy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Training status | 8 months
  Number of certified endoscopy training centers all over the world

SECONDARY OUTCOMES:
Unmet needs | 8 months
  Identifying the unmet needs for endoscopy training all over the world

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alboraie, MD, MRCP(UK), Principal Investigator — Al-Azhay University, Cairo, Egypt
Locations (13):
- Kings County Hospital Center, Brooklyn, NY, USA, Albertson, New York, United States
- Erasme Hospital, Gastroenterology Department, Université Libre de Bruxelles (ULB), Brussels, Belgium
- São Lucas Academic Hospital - Gastroclínica Cascavel, Cascavel, Brazil
- Hospital Luis Calvo Mackenna and Clínica Alemana de Santiago, Santiago, Chile
- Egypt (2):
  - Al-Azhar Univerisity, Cairo, Cairo Governorate
  - Faculty of Medicine, Zagazig University, Zagazig, Sharqia Province
- Ahvaz Imam hospital, Ahvāz, Ahvaz, Iran
- Dow university of health sciences, Civil hospital Karachi, Karachi, Pakistan
- Pomeranian Medical University, Szczecin, Poland
- Singapore General Hospital, Singapore, Singapore
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan
- Koç University Hospital, Istanbul, Istanbul, Turkey (Türkiye)
- The Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Final results will be made available but not individual participant data.

REFERENCES:
- [Result] Losowsky MS. Research, education, science, training. Work of the committees. British Society of Gastroenterology. Gut. 1987 Sep;28 Suppl(Suppl):25-6. No abstract available. PMID 3311912
- [Result] ASGE Training Committee; Adler DG, Bakis G, Coyle WJ, DeGregorio B, Dua KS, Lee LS, McHenry L Jr, Pais SA, Rajan E, Sedlack RE, Shami VM, Faulx AL. Principles of training in GI endoscopy. Gastrointest Endosc. 2012 Feb;75(2):231-5. doi: 10.1016/j.gie.2011.09.008. Epub 2011 Dec 7. No abstract available. PMID 22154419
- [Result] Rutter MD, Senore C, Bisschops R, Domagk D, Valori R, Kaminski MF, Spada C, Bretthauer M, Bennett C, Bellisario C, Minozzi S, Hassan C, Rees C, Dinis-Ribeiro M, Hucl T, Ponchon T, Aabakken L, Fockens P. The European Society of Gastrointestinal Endoscopy Quality Improvement Initiative: developing performance measures. United European Gastroenterol J. 2016 Feb;4(1):30-41. doi: 10.1177/2050640615624631. Epub 2015 Dec 17. PMID 26966520
- [Result] Xiong X, Barkun AN, Waschke K, Martel M; Canadian Gastroenterology Training Program Directors. Current status of core and advanced adult gastrointestinal endoscopy training in Canada: Survey of existing accredited programs. Can J Gastroenterol. 2013;27(5):267-72. doi: 10.1155/2013/186284. PMID 23712301
- [Result] Makmun D. Present status of endoscopy, therapeutic endoscopy and the endoscopy training system in Indonesia. Dig Endosc. 2014 Apr;26 Suppl 2:2-9. doi: 10.1111/den.12245. PMID 24750141
- [Result] Ismaila BO, Misauno MA. Gastrointestinal endoscopy in Nigeria--a prospective two year audit. Pan Afr Med J. 2013;14:22. doi: 10.11604/pamj.2013.14.22.1865. Epub 2013 Jan 15. PMID 23503686
- [Result] Watermeyer G, Van Wyk ME, Goldberg PA. Audit of provincial gastroenterology services in the Western Cape. S Afr J Surg. 2008 Aug;46(3):68-72. PMID 18807301
- See also: Survey link — https://www.surveymonkey.com/r/DS7FGXF